CLINICAL TRIAL: NCT03493074
Title: Non-invasive Peri- and Postoperative Monitoring of Endovascular Repair of Abdominal Aortic Aneurysm
Brief Title: Non-invasive Monitoring of Endovascular Repair of Abdominal Aortic Aneurysm (VBA)
Acronym: VBA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University of Technology (Other); Tampere University (Other)
Responsible Party: Sponsor
Other Study IDs: R17129
Record Dates: First submitted 2018-03-20; First posted 2018-04-10 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Cardiovascular Diseases; Abdominal Aortic Aneurysm
MeSH Terms: conditions — Cardiovascular Diseases; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Noninvasive pulse wave analysis sensor, ECG-sensor — The sensors are noninvasively attached

SUMMARY:
This study evaluates a novel noninvasive method to dynamically monitor the effect of abdominal aortic aneurysm (AAA) and endovascular treatment of AAA (EVAR) on arterial pulse wave

DETAILED DESCRIPTION:
Abdominal aortic aneurysm (AAA) develops slowly and degeneratively (increasing diameter, wall tension, thinning and decreased wall strength, altered compliance) which affects the aortic pressure and wave reflection. In 50% of cases, AAA rupture may lead to death and 50% of the remaining patients referred to hospital die. This results in high costs and preventable loss of lives. AAA can also be detected by pulse wave (PW) analysis. which could enable development of easy to use, affordable and accurate methodology for the detection of AAAs. The measurement system used in the present study is capable of wireless recording of PWs from several different locations utilizing two different sensor modalities (blood-volume related photoplethysmographic (PPG) PWs and dynamic blood pressure PWs). The objective is to study PWs in the detection of AAA and the effects of endovascular repair (EVAR) and whether adverse effects (i.e. endograft failure) can be detected. It is hypothesized that AAA and failure of the operation can be detected by PW features, especially by printed flexible sensors which will improve the usability, patient comfort and safety (hygiene). The technology could make it possible to screen AAAs at lower costs even in the municipal health centers or by the patients themselves, at similar accuracy, without skilled personnel operating the diagnostic devices and therefore improve the cost effectiveness of AAA screening resulting in significant savings, resource reallocation in the healthcare and also improved patient safety and prevention of deaths. It could also enable patient-centered, comfort follow-up for patients treated by EVAR.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been clinically examined at policlinic of vascular surgery
* The patient has been examined with computed tomography (CT) imaging
* The patient has been considered a candidate for the EVAR of the AAA

Exclusion Criteria:

* A patient has a pacemaker
* A medical doctor decides that the measurement disturbs or risks the subject's treatment process
* Subject's denial (or withdrawal)
* A patient has at least one amputated limb
* The age of the test subject candidate is less than 18 years
* A test subject candidate is not able to understand the study or is not legally competent
* A test subject candidate has Ehlers-Danlos syndrome or Marfan syndrome

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Finnish, Caucasian
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-04-08 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Pulse wave change from baseline during EVAR measured by a force sensor | 2 hours
  A force sensor node for dynamic pressure-PW measurements is utilized to detect pulse wave
Pulse wave change from baseline during EVAR measured by a optical photoplethysmographic (PPG) sensor | 2 hours
  Optical photoplethysmographic (PPG) sensor node is used for volume pulse measurements

SECONDARY OUTCOMES:
Pulse wave change from baseline after EVAR measured by a force sensor | 30 days
  A force sensor node for dynamic pressure-PW measurements is utilized to detect pulse wave
Pulse wave change from baseline after EVAR measured by a optical photoplethysmographic (PPG) sensor | 30 days
  Optical photoplethysmographic (PPG) sensor node is used for volume pulse measurements
Pulse wave change from baseline after EVAR measured by a force sensor | 12 months
  A force sensor node for dynamic pressure-PW measurements is utilized to detect pulse wave
Pulse wave change from baseline after EVAR measured by a optical | 12 months
  Optical photoplethysmographic (PPG) sensor node is used for volume pulse measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Undecided